CLINICAL TRIAL: NCT06460311
Title: Effects Of Pediatric Endurance And Limb Strengthening (PEDAL) Program With And Without Electrical Muscle Stimulation On Mobility And Gait In Children With Cerebral Palsy
Brief Title: Effects of PEDAL Program With and Without EMS On Mobility And Gait In Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR &AHS/23/0799
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; electrical muscle stimulation; cycling; gait analysis; mobility; stationary cycle
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): PEDAL and EMS
  Interventions: Other: PEDAL and EMS
- Group B (Active Comparator): PEDAL
  Interventions: Other: PEDAL

INTERVENTIONS:
Other: PEDAL and EMS — Group A will receive EMS with Stationary cycle. EMS will be given at quadricep muscles. The pads will placed vertically in the midline along the knee and the pelvis. EMS will be given at frequency = 35 to 70 Hz, pulse duration = 100 μs, pulse period = 50 ms, Intervention will be will be performed for 60 minutes for 3 times or week for 4 weeks.
  Conversely, the endurance training phase will involve securing the cycle seat while children cycle at their maximum capacity, aiming for a heart rate between 70% to 80% of their maximum. Prior to and following each session, stretching exercises targeting the calf, quadricep, and hamstring muscles will be administered, with a 10-second hold during both the warm-up and cool-down sessions. Pre and post measurements will be conducted to evaluate mobility and gait
  Arms: Group A
Other: PEDAL — In Group B, participants will exclusively receive the Pediatric Endurance and Limb Strengthening program without EMS. Similar to Group A, this program will incorporate the use of a stationary cycle. The warm-up and cool-down periods will also include a 10-second hold for each targeted muscle group. The intervention will consist of 60-minute sessions conducted three times per week over a span of four weeks.
  Pre and post-assessments of gait and mobility will be conducted using the Gait Outcomes Assessment List (GOALTM) Questionnaire and the time up and go test.
  Arms: Group B

SUMMARY:
PEDAL is a program that focuses on juvenile endurance and limb building for kids with cerebral palsy. Studying how PEDAL with and without Electrical Muscle Stimulation (EMS) affects these metrics in an effort to determine whether exercise and EMS together can improve functional outcomes for young cerebral palsy patients. This research provides important new understandings into customized therapies to improve mobility in kids with this neurological disorder. On -- participants, a randomized controlled study will be carried out. The Zunnorain Foundation in Faisalabad will provide the data through the use of a non-probability convenience sampling method. This study will involve children with cerebral palsy who are between the ages of 6 and 12 and who can understand real directions, as well as those who have fair or good selective motor control. On the other hand, children who use orthotics or take oral medications, or those who have had any surgery or implant within the last year, are not allowed to participate in this study. The 22-person sample is split into two groups. Group A will get a comprehensive intervention consisting of a stationary cycle and electrical muscle stimulation (EMS). . EMS will be applied to the quadricep muscles using specific parameters (frequency = 35 to 70 Hz, pulse duration = 100 μs, pulse period = 50 ms). There are two stages to the stationary cycle program: an endurance phase and a strengthening phase. Group B, on the other hand, will just get the pediatric endurance and limb-strengthening program. Warm-up and cool-down phases of this program include stationary cycle assistance. Each muscle is held for 10 seconds. For four weeks, each of the two groups will receive 60 minutes of treatment three times a week. Using the Gait Outcomes Assessment List (GOALTM) Questionnaire and the time up and go test, gait and mobility will be evaluated in both groups before and after the intervention.

DETAILED DESCRIPTION:
Group A (PEDAL+EMS Group)

Group A will receive EMS with Stationary cycle. EMS will be given at quadricep muscles. The pads will placed vertically in the midline along the knee and the pelvis. EMS will be given at frequency = 35 to 70 Hz, pulse duration = 100 μs, pulse period = 50 ms, Intervention will be will be performed for 60 minutes for 3 times or week for 4 weeks.

Contrastingly, the stationary cycle will be administered in two distinct phases: strengthening and endurance. During the lower extremity strengthening phase, the cycle seat will be adjusted by sliding it backward along a linear track. The resistance of the cycle will be augmented once the participant can easily complete 10 revolutions with the seat unlocked. Conversely, the endurance training phase will involve securing the cycle seat while children cycle at their maximum capacity, aiming for a heart rate between 70% to 80% of their maximum. Prior to and following each session, stretching exercises targeting the calf, quadricep, and hamstring muscles will be administered, with a 10-second hold during both the warm-up and cool-down sessions. Pre and post measurements will be conducted to evaluate mobility and gait.

Group B (PEDAL Group

ChatGPT In Group B, participants will exclusively receive the Pediatric Endurance and Limb Strengthening program without EMS. Similar to Group A, this program will incorporate the use of a stationary cycle. The warm-up and cool-down periods will also include a 10-second hold for each targeted muscle group. The intervention will consist of 60-minute sessions conducted three times per week over a span of four weeks.

Pre and post-assessments of gait and mobility will be conducted using the Gait Outcomes Assessment List (GOALTM) Questionnaire and the time up and go test.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 12 years
* Ability to follow simple verbal directions
* Good or fair selective motor control for at least one lower limb
* Ability to walk independently indoors, with or without assistive devices (Levels I-III of the Gross Motor Function

Exclusion Criteria:

* Orthopedic surgery, neurological surgery or baclofen pump implantation within the preceding 12 months
* Serial casting or new orthotics within the preceding three months
* Initiating oral medications that affect the neuromuscular system, e.g. baclofen, within the preceding three months
* Onset of physical therapy, exercise, sport activity or change in assistive devices for walking within the preceding three months
* Inability or unwillingness to maintain age appropriate behavior
* Serious medical conditions such as cardiac disease, diabetes or uncontrolled seizures
* Current participation in a fitness program that includes cardiorespiratory endurance exercise, at least one time per week

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Selective Control Assessment of Lower Extremity (SCALE) | 8 Weeks
  The SCALE tool is a clinical assessment instrument made for medical practitioners to test selective voluntary motor control (SVMC) without the use of specialized equipment and in 15 minutes. Bilateral examinations of the hip, knee, ankle, subtalar, and toe joints are carried out. Its scoring range is from 0 to 2 where 2 shows normal and 0 shows unable. The maximum score of each leg is 10. The findings demonstrated high reliability and validity ranging from 0.88 to 0.91
o Timed Up and Go Test Time Up And Go Test o Timed Up and Go Test o Timed Up and Go Test o Timed Up and Go Test | 8 Weeks
  Time up and go test is used to assess person's static and dynamic mobility. It includes the time person takes to stand, walk, turn, walk and sit down again. Its assessment is done in seconds. It is a very valid and reliable tool 0.97 and 0.99
Gait Outcomes Assessment List (GOALTM) Questionnaire Parent Version | 8 Weeks
  This is questionnaire is used to assess functional mobility and gait among childrens of cerebral palsy. This is a 48 item questionnaire with seven domains. Its maximum score is 100. Higher score show higher function. It is a valid and reliable tool. It has a reliability of 0.92 and validity of 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Aslam, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitrikas K, Dalton H, Breish D. Cerebral Palsy: An Overview. Am Fam Physician. 2020 Feb 15;101(4):213-220. PMID 32053326